CLINICAL TRIAL: NCT04152655
Title: A Study of Efficacy and Safety of Idebenone Vs. Placebo in Prodromal Parkinson Disease (SEASEiPPD)
Brief Title: A Study of Efficacy and Safety of Idebenone Vs. Placebo in Prodromal Parkinson Disease
Acronym: SEASEiPPD
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Due to COVID-19 pandemic, in-hospital polysomnography and visits were infeasible.
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Peking Union Medical College Hospital (Other); Beijing Hospital (Other Government); Beijing Tiantan Hospital (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Jiangsu Province Nanjing Brain Hospital (Other); The First Affiliated Hospital of Anhui Medical University (Other); Huashan Hospital (Other); Tongji Hospital (Other); Second Affiliated Hospital of Soochow University (Other); Guizhou Medical University (Other); The First Affiliated Hospital of Guangzhou Medical University (Other); Peking University Shenzhen Hospital (Other); West China Hospital (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Sir Run Run Shaw Hospital (Other); The Affiliated Hospital of Hangzhou Normal University (Other); The First Affiliated Hospital of Dalian Medical University (Other); Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019-278
Record Dates: First submitted 2019-10-07; First posted 2019-11-05 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2021-07

CONDITIONS: REM Sleep Behavior Disorder; Parkinson Disease
MeSH Terms: conditions — REM Sleep Behavior Disorder; Parkinson Disease | interventions — idebenone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1: idebenone (Active Comparator): Oral 30 mg fixed dose three times a day x 24-months (90 mg total / day) with assessments @ baseline, 3 month, 6 month, 12 month, 15 month, 18 month, 21 month and 24 months
  Interventions: Drug: Idebenone
- Group 2: placebo (Placebo Comparator): Oral placebo three times a day x 24-months with assessments @ baseline, 3 month, 6 month, 12 month, 15 month, 18 month, 21 month and 24 months
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Idebenone — 30mg tablets three times a day
  Other Names: Coenzyme Q10 analogue
  Arms: Group 1: idebenone
Drug: Placebo oral tablet — placebo tablets three times a day
  Arms: Group 2: placebo

SUMMARY:
To investigate whether 24 months of idebenone may reduce the progression from Prodromal Parkinson disease (PPD) to Parkinson disease (PD).

DETAILED DESCRIPTION:
Number of people suffered from Parkinson disease (PD) is increasing every year. Contemporary medication has little neuroprotective effect, which may due to delayed treatment as over 50% neurons have lost when clinical diagnosed PD emerges. The concept of Prodromal Parkinson disease (PPD) is emphasized as it has become evident that there are several risk and clinical markers may occur years before the cardinal motor symptoms which allow clinical diagnosis. Rapid eye movement (REM) sleep behavior disorder and olfactory dysfunction are the most common PPD, and more than one third of patients may progress to PD and other neurodegenerative diseases. Mitochondrial injury is one of the pathogenesis of PD. Thus we design this trial to investigate whether idebenone, potent coenzyme Q10 analogue, could protect PPD develops into PD.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are voluntary to participate and have signed informed consent
* Diagnosed as Rapid Eye movement (REM) Sleep Behavior Disorder by polysomnography

Exclusion Criteria:

* Subjects are pregnant, breastfeeding, or want to get pregnant or breastfeeding in 2 years
* Subjects have history of allergy to idebenone
* Difficulty to communicate
* Suffering from neurodegenerative diseases
* Having obvious brain imaging abnormalities (eg. severe brain atrophy, malformation, softening lesions, cerebrovascular disease, intracranial occupancy, giant large benign lesions, etc.)
* Having severe mental illness (eg. schizophrenia, manic depression, and severe depression)
* Long-term use of clonidine, dopamine antagonists, and serotonin reuptake inhibitors
* Suffering from other severe medical conditions
* Having difficulty in moving and are unable to come to the hospital
* Having claustrophobia
* Having contraindications to MRI tests
* Having history of olfactory disorders greater than 10 years
* Having history of color vision disorders greater than 10 years
* Life expectancy less than 2 years
* Having other situations which researchers consider is inappropriate to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Clinical diagnosis of parkinson disease | 24 months
  based on Movement Disorder Society (MDS) Research Criteria for Prodromal Parkinson's Disease in 2015

SECONDARY OUTCOMES:
Dopamine transporter positron emission tomography (DAT-PET) change | 12 month and 24 month
  diminishment of striatal DAT-PET
Quantitative motor testing change | 24 months
  Unified Parkinson Disease Rating Scale, Part III

CONTACTS AND LOCATIONS:
Overall Officials: Baorong Zhang, MD, Study Chair — Second Affiliated Hospital of Zhejiang University School of Medicine
Locations (1):
- Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes